CLINICAL TRIAL: NCT00803556
Title: Phase 1 Clinical Trial of the Combination of Intravenous Alvespimycin (KOS-1022), Trastuzumab With or Without Paclitaxel
Brief Title: Clinical Trial of the Combination of Intravenous Alvespimycin (KOS-1022), Trastuzumab With or Without Paclitaxel in Patients With Advanced Solid Tumor Malignancies or Her2 Positive Metastatic Breast Cancer Who Have Previously Failed Trastuzumab Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA201-001; KDG 132
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Solid Tumor; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 17-(dimethylaminoethylamino)-17-demethoxygeldanamycin; Trastuzumab; Paclitaxel; BMS 181339

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Patients whose last dose is > 21 days prior to first dose of Trastuzumab on study. First infusion: 90 mins for 4 mg/kg loading dose of trastuzumab followed by 60 min infusion of alvespimycin. Subsequent infusions weekly 30 mins for 2 mg/kg trastuzumab followed by 60 min infusion of alvespimycin
  Patients whose last dose is < 21 days prior to first dose of Trastuzumab on study. All infusions: 30 mins for 2 mg/kg trastuzumab followed by 60 min infusion of alvespimycin
  Interventions: Drug: Alvespimycin; Drug: Trastuzumab
- Arm 2 (Experimental): Patients whose last dose is > 21 days prior to first dose of Trastuzumab on study. First infusion: 90 mins for 4 mg/kg loading dose of trastuzumab followed by 60 min infusion of paclitaxel and 60 min of infusion of alvespimycin. Subsequent infusions weekly 30 mins for 2 mg/kg trastuzumab followed by 60 min infusion of paclitaxel and 60 min infusion of alvespimycin
  Patients whose last dose is < 21 days prior to first dose of Trastuzumab on study. All infusions: 30 mins for 2 mg/kg trastuzumab followed by 60 min infusion of paclitaxel and 60 min infusion of alvespimycin. Subsequent infusions weekly 30 mins for 2 mg/kg trastuzumab followed by 60 min infusion of paclitaxel and 60 min infusion of alvespimycin
  Interventions: Drug: Alvespimycin; Drug: Trastuzumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Alvespimycin — Solution, IV, 60-100 mg/m2, weekly until disease progression or DLT
  Other Names: BMS-826476
Drug: Trastuzumab — Solution, IV, 2-4 mg/kg, weekly until disease progression or DLT
  Other Names: Herceptin; BMS-722782
Drug: Paclitaxel — Solution, IV, 60-90 mg/m2, weekly until disease progression or DLT
  Other Names: Taxol; BMS-181339
  Arms: Arm 2

SUMMARY:
To determine the Maximally Tolerable Dose (MTD) of KOS-1022 when administered weekly in combination with trastuzumab or in combination with trastuzumab and paclitaxel to patients with advanced solid tumor malignancies

ELIGIBILITY:
Inclusion Criteria:

* KPS performance status >= 70%
* Schedule A: all patients must have a histologically confirmed solid tumor malignancy. Schedule B: patients must have metastatic breast cancer with Her2 amplification by FISH or 3+ Her2 overexpression by immunohistochemistry ("IHC"). Patients are not required to have measurable disease for this investigation. Disease must be assessed within 28 days prior to treatment initiation
* All Adverse Events of any prior chemotherapy, surgery, or radiotherapy, must have resolved to NCI CTCAE (v. 3.0) Grade <= 2 (except for alopecia)
* The following laboratory results, within 10 days of KOS-1022 administration:

  * Hemoglobin >= 8.5 g/dL
  * Absolute neutrophils count >= 1.5 x 10*9* /L
  * Platelet count >= 75 x 10*9*/L
  * Serum bilirubin <= 2 x ULN
  * AST and ALT <= 2.5 x ULN
  * Serum creatinine <= 2 x ULN

Exclusion Criteria:

* Documented hypersensitivity reaction of CTCAE Grade >= 3 to prior therapy containing trastuzumab
* Pregnant or breast-feeding women. Male patients must be surgically sterile or agree to use an acceptable method of contraception
* Known active CNS metastases
* Administration of any other chemotherapy, biological, immunotherapy or investigational agent (therapeutic or diagnostic) within 14 days prior to receipt of study medication. Patients should be 6 weeks from last dose of nitrosourea
* Patients with Grade 2 or higher dyspnea at rest on room air; patients with other clinically significant pulmonary co-morbidity(s) that might predispose the patient to pulmonary toxicity
* Moderately severe dry eye
* Prior pulmonary toxic chemotherapy (e.g, bleomycin or carmustine)
* Congestive heart failure, or a left ventricular ejection fraction (LVEF)
* Any medical conditions that, in the Investigator's opinion, would impose excessive risk to the patient
* Patients with previous malignancies unless free of recurrence for at least 5 years except cured basal cell carcinoma of the skin, carcinoma-in-situ of either the uterine cervix or urinary bladder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Number of Dose Limiting Toxicities | During Cycle 1 (4-weeks in duration)

SECONDARY OUTCOMES:
Summary of Adverse Events, Serious Adverse Events, Deaths and Discontinuations due to Adverse Events | Weekly
Summary of Clinical Laboratory Abnormalities | Weekly
AUC of KOS-1022 and its metabolites | Week 1 and Week 4: pretreatment, 30 and 55 minutes after start of infusion, 5, 15, 30 minutes and 1, 2, 4, 6, 24, 72 hours post-infusion; Weeks 2 and 3: pre-infusion
Cmax of KOS-1022 and its metabolites | Week 1 and Week 4: pretreatment, 30 and 55 minutes after start of infusion, 5, 15, 30 minutes and 1, 2, 4, 6, 24, 72 hours post-infusion; Weeks 2 and 3: pre-infusion
T-Half of KOS-1022 and its metabolites | Week 1 and Week 4: pretreatment, 30 and 55 minutes after start of infusion, 5, 15, 30 minutes and 1, 2, 4, 6, 24, 72 hours post-infusion; Weeks 2 and 3: pre-infusion
Expression of Hsp90-client proteins in peripheral blood lymphocytes | Pretreatment, 4 hours following the Day 1 KOS-1022 infusion, Day 2, Day 4; pretreatment samples Weeks 2 and 3; pretreatment, 4 hours following the Day 22 KOS-1022 infusion, Day 23, Day 25
Tumor response as assessed by RECIST criteria first after two cycles of therapy | For patients with measurable disease, response will be assessed by RECIST criteria first after two cycles of therapy (8 weeks in patients having no delay in the schedule of administration)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx